CLINICAL TRIAL: NCT00123019
Title: Overweight and Obesity Control in Worksites
Brief Title: Work, Weight, and Wellness Program: The 3W Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Thomas M. Vogt, MD, MPH, Kaiser Permanente Center for Health Research, Hawaii
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 230; R01HL079505 (NIH); NCT00119808 (obsolete NCT alias)
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2009-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity | interventions — Exercise; Diet

ARMS (2):
- 1 (Active Comparator): Minimal intervention; annual weight/waist assessment, questionnaire, and advice
  Interventions: Behavioral: Exercise and diet; Behavioral: Level 1
- 2 (Experimental): Intensive intervention. All arm 1 activities plus ongoing environmental and group interventions in worksite for two years.
  Interventions: Behavioral: Diet, Weight Reducing; Behavioral: Level 2

INTERVENTIONS:
Behavioral: Exercise and diet — Advice and measurement only
  Arms: 1
Behavioral: Diet, Weight Reducing — Measurement, advice, environmental and behavioral group interventions
  Arms: 2
Behavioral: Level 1 — Annual assessment of weight and waist circumference, questionnaire on work, health issues, advice on diet, physical activity and other health issues.
  Arms: 1
Behavioral: Level 2 — All Level 1 activities plus ongoing environmental interventions in worksite and weight management groups in worksite over a 24 month period.
  Arms: 2

SUMMARY:
The purpose of this study is to increase physical activity, improve diet, and reduce obesity of hotel employees.

DETAILED DESCRIPTION:
BACKGROUND:

In Hawaii, as in many other states, tourism is a large industry. Most hotel jobs require little education or training, and hotels employ large numbers of persons and immigrants with low socioeconomic status. Hawaii, with the world's most ethnically diverse population, has high rates of obesity and diabetes, particularly among those of Polynesian ancestry (about 20-22% of the population). This study will include a comprehensive lifestyle change program delivered through worksites in partnership with a large health care system.

DESIGN NARRATIVE:

Thirty-one hotels employing 11,000 persons on the island of Oahu are pair-matched. One member of each pair is assigned to a high intensity intervention and the other to a low intensity intervention. Both interventions are intended to reduce BMI through an emphasis on a healthy diet and increased physical activity. All employees are assessed annually for three consecutive years. The assessment includes a survey on lifestyle habits, stage of change, and attitudes toward weight, as well as measurement of BMI. The high intensity intervention hotels receive the following: 1) environmental changes to support lifestyle change and obesity control; 2) worksite based groups that offer state-of-the-art behavioral interventions; and 3) after-hours "Re-Invent Yourself" groups designed for persons who want to lose at least 25 pounds and are highly committed to doing it. These interventions incorporate all the elements that produce sustained weight loss and an innovative decision tutorial based on decision theory. The primary outcome is the mean difference between hotels in the high intensity and low intensity interventions in change in BMI from baseline to 12 and 24 months. Secondary outcomes address effects of the intervention on ethnic and occupational subgroups stage of change, absentee days, and worker compensation claims.

ELIGIBILITY:
Inclusion Criteria:

* Employed at the hotel

Exclusion Criteria:

* Unable to read English, Korean, or Chinese

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6100 (Estimated)
Dates: Start 2004-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Change in BMI | Measured at Months 12 and 24

SECONDARY OUTCOMES:
Effects of the intervention on ethnic and occupational subgroups, stage of change, and other issues | Measured at Months 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Vogt, MD, MPH, Study Chair — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Hawaii, Honolulu, Hawaii, United States